CLINICAL TRIAL: NCT02102789
Title: Systemic Chemotherapy With or Without Hepatic Arterial Infusion With Floxuridine in Patients With Initially Unresectable Colorectal Liver Metastasis: A Prospective, Randomised, Controlled Study
Brief Title: A Study of Systemic Chemotherapy With/Without HAI in Patients With Initially Unresectable Colorectal Liver Metastasis
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhong Li (Other)
Responsible Party: Sponsor-Investigator, Yuhong Li, MD, Ph D, Sun Yat-sen University
Organization: Sun Yat-sen University (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Frozen-2
Record Dates: First submitted 2014-03-31; First posted 2014-04-03 (Estimated); Last update posted 2024-03-04 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Oxaliplatin; Leucovorin; Fluorouracil; Floxuridine; Dexamethasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Systemic chemotherapy (Experimental): Patients will receive mFOLFOX6 every 28 days: Oxaliplatin 85 mg/m2 IV over 3 hours on Day 1, 15; Leucovorin (l-LV) 200mg/m2 IV over 2 hours on Day 1, 15; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion on Day 1, 15.
  Interventions: Drug: mFOLFOX6
- Systemic chemotherapy combined with HAI (Experimental): Patients will receive mFOLFOX6+HAI every 28 days: Oxaliplatin 85 mg/m2 IV over 3 hours on Day 1, 15; Leucovorin (l-LV) 200mg/m2 IV over 2 hours on Day 1, 15; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion on Day 1, 15. 0.12 mg/kg/day floxuridine (FUDR) and 25 mg dexamethasone in normal saline to a total volume of 300 ml will be administered through the HAI pump.
  This will be repeated on Day 1 of each 28-day cycle. FUDR will be administered through a 14-day continuous infusion with the HAI pump.
  Interventions: Drug: mFOLFOX6; Drug: HAI

INTERVENTIONS:
Drug: mFOLFOX6 — Patients will receive mFOLFOX6 every 28 days: Oxaliplatin 85 mg/m2 IV over 3 hours on Day 1, 15; Leucovorin (l-LV) 200mg/m2 IV over 2 hours on Day 1, 15; followed by 5-Fluorouracil 2.4 g/m2 for 46 hours continuous infusion on Day 1, 15.
  Other Names: Oxaliplatin; Leucovorin; 5-fluorouracil
Drug: HAI — Patients will receive HAI every 28 days: 0.12 mg/kg/day floxuridine (FUDR) and 25 mg dexamethasone in normal saline to a total volume of 300 ml will be administered through the HAI pump.
  This will be repeated on Day 1 of each 28 day cycle. FUDR administration will be a 14-day continuous infusion using the HAI pump.
  Other Names: floxuridine (FUDR); dexamethasone
  Arms: Systemic chemotherapy combined with HAI

SUMMARY:
The primary objective of this study is to determine whether systemic chemotherapy combined with hepatic arterial infusion with floxuridine and dexamethasone can increase the complete resection rate (R0) and improve the overall survival in patients with initially unresectable colorectal liver metastasis.

DETAILED DESCRIPTION:
Recent studies and our experience have proved the efficacy and safety of systemic chemotherapy combined with hepatic arterial infusion (HAI) with floxuridine and dexamethasone in patients with initially unresectable colorectal liver metastasis. However, most of them are retrospective studies, phase I or II clinical researches, which could not provide high-level evidence. Therefore, we designed this study to determine whether systemic chemotherapy combined with HAI can increase the complete resection rate (R0) and improve the overall survival in patients with initially unresectable colorectal liver metastasis.

ELIGIBILITY:
Inclusion Criteria:

* Age: 18-70 years old
* Histologically confirmed colorectal adenocarcinoma
* Radiologically or pathologically confirmed diagnosis of colorectal liver metastasis
* Initially unresectable colorectal liver metastasis confirmed by the multidisciplinary team (MDT)
* With no prior treatment for liver metastasis, including chemotherapy, operation, radiotherapy, transcatheter hepatic arterial chemoembolization (TACE) and targeted therapy
* Without extra-hepatic metastasis confirmed by CT, MRI or PET/CT (if necessary) scanning
* With adequate bone marrow function: platelets ≥ 90 x 109/L; white blood cells ≥ 3×109/L; absolute neutrophil count (ANC) ≥ 1.5 x 109/L
* Serum bilirubin ≤ 1.5 x ULN, AST and ALT ≤ 5 x ULN
* Patient has no ascites and with adequate blood coagulation function, albumin ≥ 35 g/L
* Grade A level of Child-Push Liver Function
* Creatinine ≤ 1× ULN, or Calculated Creatinine Clearance >50ml/min （Cockcroft-Gault Equation）
* ECOG performance status of 0-2
* Life expectancy ≥ 3 months
* Not appropriate for anti-EGFR or any other targeted therapy (with KRAS mutation or could not afford it)
* Patients have provided a signed Informed Consent Form
* With good compliance

Exclusion Criteria:

* With any extra-hepatic metastasis and/or primary tumor recurrence
* Severe arterial embolism or ascites
* With hemorrhagic tendency or coagulation disorders
* Hypertensive crisis or hypertensive encephalopathy
* Severe and uncontrolled systemic complications such as infections or diabetes
* Serious cardiovascular diseases such as cerebrovascular accident (within 6 months before enrollment), myocardial infarction (within 6 months before enrollment), uncontrolled hypertension even with appropriate drug intervention, unstable angina pectoris, congestive heart failure (NYHA 2-4 degree), arrhythmia that needs medication intervention
* Patient who has suffered from central nervous system diseases such as primary brain tumor, uncontrolled epilepsy even with standard treatment, any brain metastasis or stroke
* Patient who has a concurrent malignancy or has a malignancy within 5 years before study enrollment, (with the exception of radically resected skin basal cell carcinoma or cervical carcinoma in situ)
* Patient who has received any investigational antineoplastic agent within 28 days before the enrollment
* Any residual toxicity from prior chemotherapy (with the exception of alopecia), such as grade 2 or more sensory peripheral neuropathy (NCI CTC v3.0), oxaliplatin-based regimen will not be considered
* Patient who is allergic to oxaliplatin, leucovorin, 5-Fluorouracil, floxuridine or dexamethasone
* Pregnant or lactating women
* Patient who does not use or refuses to take any appropriate contraceptive measures (intrauterine contraceptive ring, barrier contraception combined with spermicidal gel or sterilization operation), including women of childbearing age (within 2 years after the last menstrual period) and men who are with possible fertility
* Unable or unwilling to comply with the research plan
* The existence of any other disease, dysfunction caused by metastatic lesions, or suspicious disease found on the regular examination, which indicating contraindications to the use of study drugs or may bring high risks of treatment related complications

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 142 (Estimated)
Dates: Start 2014-03; Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Complete resection rates (R0 resection rates) (defined as no macroscopic or microscopic residual tumor) of both arms | Up to 2-4 months

SECONDARY OUTCOMES:
Overall response rates (ORR) of both arms | Up to 4-8 monthes
R1 resection rates (with microscopic residual tumor) of both arms | Up to 2-4 monthes
Specific R0/R1 resection plus radiofrequency ablation rates of both arms | Up to 2-4 monthes
Recurrence-free survival (RFS) of both arms | Up to 5 years
  Time to recurrence or death
5 year cancer specific survival rate of the whole population | Up to 5 years
Progression free survival(PFS) of both arms | From the date of first drug administration until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 monthes
Overall survival (OS) of both arms | From the date of first drug administration until the date of death, assessed up to 5 years
Number of participants with surgical complications, AES and SAEs as a measure of safety | Each follow up visit, assessed up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Yu-hong Li, MD, Ph D, Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China